CLINICAL TRIAL: NCT03084146
Title: The Role of Food Sensitivity in Psoriasis: a 12-week Prospective Correlational Study of the Impact of an Individualized Elimination Diet on Disease Severity
Brief Title: The Role of Food Sensitivity in Psoriasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Yolanda Rosi Helfrich, Director Program for Clinical Research In Dermatology, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Derm 685/HUM00115672
Record Dates: First submitted 2017-02-23; First posted 2017-03-20 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Elimination Diets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psoriasis (Experimental): Psoriasis patients will be placed on an individualized 12-week elimination diet
  Interventions: Other: 12-week elimination diet
- Healthy Control (No Intervention): Healthy Control patients will receive no intervention

INTERVENTIONS:
Other: 12-week elimination diet — individualized 12-week elimination diet based on the 4 most reactive foods +/- a gluten-free diet if there is detection of positive anti- tissue transglutaminase (tTG) IgG and IgA and anti-deamidated gliadin peptide (DGP) IgG and IgA
  Arms: Psoriasis

SUMMARY:
Psoriasis is a common chronic skin disorder that affects over 4 million people. There is no cure for psoriasis and treatment is directed at controlling patients' symptoms. The purpose of this study is to determine whether psoriasis patients are more likely to have food sensitivities than those patients without psoriasis. We will also determine if eliminating certain foods from the diet results in a change in psoriasis symptoms.

DETAILED DESCRIPTION:
Purpose: To determine the role of food sensitivity in psoriasis and assess the clinical response of an individualized elimination diet on psoriasis.

Design: Up to 50 volunteers with psoriasis and 20 age- and sex-matched controls will be recruited for a 12-week prospective correlational study.

Methods: Venous blood samples for the detection of antibodies against food antigens will be collected and individualized elimination diets will be designed based on the most reactive food antigens.

Assessments: Clinical assessments of objective and subjective parameters will be measured using Psoriasis Area and Severity Index (PASI), Static Physicians Global Assessment (sPGA), Dermatology Life Quality Index (DLQI), and Itch Numeric Rating Scale (Itch NRS).

Objectives: The primary objectives are to determine whether psoriasis patients are more likely to have food sensitivities and assess the clinical response of a 12-week elimination diet on psoriasis.

ELIGIBILITY:
Inclusion criteria:

* Male or female subjects, 12 years of age or older.
* Good general health.
* Willingness and ability to follow the protocol.
* Signed Informed Consent Form, written and witnessed.
* Psoriatic group only: Chronic plaque psoriasis (patients must have diagnosis for at least 6 months) or guttate psoriasis involving 2 % or greater total body surface area or 2 plaques, each measuring > 8 cm2.
* Psoriatic group only: Psoriasis is untreated (as defined in Exclusion criteria 4) or subject has been on a stable topical or systemic treatment with no dose alteration or regimen alteration for >12 months.

Exclusion criteria:

* History of drug-induced psoriasis or pustular psoriasis.
* Moderate or severe psoriasis warranting systemic immunosuppression or inpatient admission.
* Pregnant, lactating, history of diabetes mellitus, thyroid disease or inflammatory bowel disease.
* Psoriatic group only: Use of biologic treatment for psoriasis within 3 months of baseline, use of systemic immunosuppressive treatment for psoriasis within 4 weeks of baseline, or use of topical treatment for psoriasis within 2 weeks.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2023-10-22 (Actual); Study Completion 2023-10-22 (Actual)

PRIMARY OUTCOMES:
IgG4 Antibodies | 12 weeks
  IgG4 Antibodies against Eliminated Food Antigens in Psoriasis Patients vs. Controls
IgE Antibodies | 12 weeks
  IgE Antibodies against Eliminated Food Antigens in Psoriasis Patients vs. Controls
Anti-Tissue Transglutaminase (tTG) IgG | 12 weeks
  Anti-Tissue Transglutaminase (tTG) IgG Change from Baseline in Psoriasis Patients vs. Controls
Anti-Tissue Transglutaminase (tTG) IgA | 12 weeks
  Anti-Tissue Transglutaminase (tTG) IgA Change from Baseline in Psoriasis Patients vs. Controls
Anti-Deamidated Gliadin Peptide (DGP) IgG | 12 weeks
  Anti-Deamidated Gliadin Peptide (DGP) IgG Change from Baseline in Psoriasis Patients vs. Controls
Anti-Deamidated Gliadin Peptide (DGP) IgA | 12 weeks
  Anti-Deamidated Gliadin Peptide (DGP) IgA Change from Baseline in Psoriasis Patients vs. Controls

SECONDARY OUTCOMES:
IgG4 Antibodies in Subset | 12 weeks
  IgG4 Antibodies against Eliminated Food Antigens in Subset of Psoriasis Patients with positive test result who participated in dietary elimination intervention
IgE Antibodies in Subset | 12 weeks
  IgE Antibodies against Eliminated Food Antigens in Subset of Psoriasis Patients with positive test result who participated in dietary elimination intervention
Anti-Tissue Transglutaminase (tTG) IgG in Subset | 12 weeks
  Anti-Tissue Transglutaminase (tTG) IgG in Subset of Psoriasis Patients with positive test result who participated in dietary elimination intervention
Anti-Tissue Transglutaminase (tTG) IgA in Subset | 12 weeks
  Anti-Tissue Transglutaminase (tTG) IgA in Subset of Psoriasis Patients with positive test result who participated in dietary elimination intervention
Anti-Deamidated Gliadin Peptide (DGP) IgG in Subset | 12 weeks
  Anti-Deamidated Gliadin Peptide (DGP) IgG in Subset of Psoriasis Patients with positive test result who participated in dietary elimination intervention
Anti-Deamidated Gliadin Peptide (DGP) IgA in Subset | 12 weeks
  Anti-Deamidated Gliadin Peptide (DGP) IgA in Subset of Psoriasis Patients with positive test result who participated in dietary elimination intervention

CONTACTS AND LOCATIONS:
Overall Officials: Yolanda Helfrich, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Department of Dermatology, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No